CLINICAL TRIAL: NCT07003178
Title: An Early Clinical Study to Evaluate the Safety and Clinical Efficacy of STR-P004 in Subjects With Relapsed/Refractory CD19-Positive B-Lymphocytic Non-Hodgkin's Lymphoma
Brief Title: A Study to Evaluate the Safety and Clinical Efficacy of STR-P004
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Starna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Starna Therapeutics P004
Record Dates: First submitted 2025-05-19; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose1 (Experimental): STR-P004 Dose1 IV
  Interventions: Drug: STR-P004
- Dose2 (Experimental): STR-P004 Dose2 IV
  Interventions: Drug: STR-P004
- Dose 3 (Experimental): STR-P004 Dose3 IV
  Interventions: Drug: STR-P004
- Dose4 (Experimental): STR-P004 Dose4 IV
  Interventions: Drug: STR-P004
- Dose5 (Experimental): STR-P004 Dose5 IV
  Interventions: Drug: STR-P004

INTERVENTIONS:
Drug: STR-P004 — An in vivo CART drug administered intravenously

SUMMARY:
This study is a single-arm, single-center, open-label, multiple-dose, dose-escalation early clinical study aimed at evaluating the safety, tolerability, and pharmacokinetic profile of STR-P004 in subjects with relapsed/refractory CD19-positive B-cell non-Hodgkin lymphoma, and preliminarily observing its antitumor activity.

DETAILED DESCRIPTION:
This study employs a dose-escalation approach combining "accelerated titration" and "traditional 3+3". Within the dose range of xxmg/kg to xxxmg/kg, five dose-escalation cohorts are planned. The escalation follows a modified Fibonacci sequence (i.e., 2, 1.67, 1.5, 1.4, 1.33, 1.33 …… 1.33-fold increments). A faster escalation rate is used in the early phase to minimize patient exposure to ineffective doses and rapidly reach the predicted effective dose range, after which the escalation rate is reduced to ensure safety and explore efficacy.

This study plans to enroll adult patients with B-cell non-Hodgkin's lymphoma (NHL). Enrolled patients will receive STR-P004 at the corresponding dose via intravenous infusion. Patients will receive weekly treatment doses starting from D1 for 4 consecutive weeks (D1, D8, D15, D22), with each 4-week period constituting a treatment cycle. Based on preliminary treatment results from Cycle 1, the investigator will decide whether to proceed with subsequent cycles, which will follow the same regimen as Cycle 1. The DLT observation period is 28 days (i.e., D1 to D28). If no DLT occurs or if no Grade ≥2 AE judged by the investigator to be related to the study drug and medically significant is observed, patients will be enrolled into the next dose group after the 28-day DLT observation period for the previous dose group is ended. During the accelerated titration phase, if a DLT or any Grade ≥2 AE judged by the investigator to be related to the study drug and medically significant occurs within 28 days, enrollment will switch to the "3+3" pattern.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsed/refractory CD19-positive B-cell non-Hodgkin's lymphoma:

  1. Age ≥18 years, regardless of gender;
  2. Life expectancy >12 weeks;
  3. ECOG score of 0-2;
  4. Diagnosis of B-cell non-Hodgkin's lymphoma confirmed by cytology or histopathology according to WHO 2016 criteria, including: diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL), and high-grade B-cell lymphoma (HGBCL);
  5. Pathologically confirmed B-cell non-Hodgkin's lymphoma meeting one of the following conditions:

     1. Relapsed/refractory B-cell non-Hodgkin's lymphoma with the best response of SD or PD after receiving at least two lines of adequate therapy, the best response of PD during or after the last line of treatment, or the best response of SD after receiving at least two cycles of the last line of treatment;
     2. For relapse or PD within 12 months after autologous stem cell transplantation (ASCT) for B-cell non-Hodgkin's lymphoma, if salvage therapy is administered, no response (SD/PD) to the last treatment is required; for relapse or PD more than 12 months after ASCT, salvage therapy is needed, and no response (SD/PD) to the last treatment is required;
  6. Hemoglobin ≥80 g/L, neutrophils ≥1.0 × 109/L, platelets ≥75 × 109/L;
  7. At least one measurable tumor lesion according to the 2014 Lugano response criteria;
  8. Hepatic and renal function, as well as cardiopulmonary function, meet the following requirements:

     1. Serum creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/min (calculated by the Cockcroft-Gault formula);
     2. Ejection fraction >50%, with no clinically significant pericardial effusion or pleural effusion detected;
     3. Baseline oxygen saturation >92%;
     4. Total bilirubin ≤1.5 × ULN (≤5 × ULN for Gilbert syndrome);
     5. ALT and AST ≤3 × ULN (≤5 × ULN for patients with liver metastases).
  9. Capable of understanding the study and having signed the informed consent form.

Exclusion Criteria:

* Subjects meeting any of the following conditions will not be eligible for participation:

  1. History of malignancies other than diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL), or high-grade B-cell lymphoma (HGBCL) within 5 years prior to screening, except for adequately treated cervix carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, or thyroid cancer after radical surgery;
  2. Presence of any of the following high-risk factors: sum of product of diameters (SPD) of lesions (all measurable lesions ≥1.5 cm in the longest diameter) ≥100 cm; bulky disease (single lesion ≥10 cm); lesions located in the pharynx or trachea with pressure symptom; lesions adjacent to critical hollow organs such as the gastrointestinal tract or bile ducts, where enlargement may press or invade surrounding organs and impair their functions;
  3. Subjects who have not completed a washout period of at least 5 half-lives since their last anticancer therapy (including I/O therapy) prior to the first dose of study treatment; for anticancer therapies with a half-life >5 days, a washout period >14 days is acceptable; or participation in any other clinical study within 4 weeks prior to the first treatment;
  4. Any of the following conditions: positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg); positive for hepatitis B e antibody (HBe-Ab) with HBV-DNA copy number above the lower limit of detection; positive for hepatitis C antibody (HCV-Ab); positive for anti-Treponema pallidum antibody (TP-Ab); positive for human immunodeficiency virus (HIV) antibody; EBV-DNA or CMV-DNA copy number above the lower limit of detection;
  5. Any unstable systemic disease, including but not limited to active infection (except for local infections), unstable angina, cerebrovascular accident or transient ischemic attack (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] class ≥III), severe arrhythmia requiring medication, or hepatic, renal, or metabolic disorders;
  6. Any uncontrolled active condition that may interfere with study participation;
  7. Any condition deemed by the investigator to compromise subject safety or interfere with the study objective;
  8. Pregnant or breastfeeding women, or subjects who plan to become pregnant during the treatment period or within 1 year after treatment completion, or male subjects whose partners plan to become pregnant within 1 year after cell infusion;
  9. Subjects receiving systemic corticosteroid therapy within 14 days prior to enrollment and judged by the investigator to require long-term use of systemic corticosteroid during treatment (excluding inhaled or topical use);
  10. Presence of central nervous system or brain metastasis symptoms or receiving treatment for central nervous system or brain metastasis (radiotherapy, surgery, or other therapy) within 3 months prior to enrollment;
  11. Subjects with conditions that impair their ability to provide written informed consent or comply with study procedures, or those unwilling or unable to adhere to study requirements.
  12. Subjects deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
In accordance with the (US) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and the ASTCT consensus. The incidence of DLT events in this trial. | 24 months
  DLTs in this trial are defined as dose-escalation phase, toxic reactions related to the study drug (including definitely related, probably related, and possibly related) that occur from the time of first receipt of STR-P004 IV infusion to the end of the first treatment cycle (i.e., D1~ D28), and primarily include hematologic and non-hematologic toxicities.
  >
  Hematologic DLT:
  - Grade 4 neutropenia does not return to ≤ grade 2 or baseline status within 28 days of G-CSF (granulocyte colony-stimulating factor) treatment and excludes involvement/infiltration due to the disease itself;
  - Grade 4 thrombocytopenia that does not return to grade ≤2 or baseline status within 28 days of rhTPO/TPO-RA (recombinant human thrombopoietin and thro

CONTACTS AND LOCATIONS:
Locations (1):
- Starna, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No